CLINICAL TRIAL: NCT05863624
Title: Postoperative Pain and Recurrences After Totally Extraperitoneal Endoscopic (TEP) vs. Lichtenstein Hernioplasty in Female Inguinal Hernia Repair: a Prospective Randomized Multi-center Study
Brief Title: Open and Endoscopic Technique in Female Inguinal Hernia Repair. FemaleHernia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Päijänne Tavastia Central Hospital (Other); North Karelia Central Hospital (Other); Jyväskylä Central Hospital (Other); Mikkeli Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5200667
Record Dates: First submitted 2023-04-17; First posted 2023-05-18 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized follow-up study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open hernioplasty (Experimental): Open Lichtenstein hernia repair
  Interventions: Procedure: Open hernioplasty
- TEP hernioplasty (Active Comparator): totally endoscopic hernia repair (TEP)
  Interventions: Procedure: TEP hernioplasty

INTERVENTIONS:
Procedure: Open hernioplasty — Inguinal hernia is operated using open surgery
  Other Names: Open Lichtenstein hernia repair
  Arms: Open hernioplasty
Procedure: TEP hernioplasty — Inguinal hernia is operated using laparoendoscopic technique
  Other Names: totally endoscopic hernia repair (TEP)
  Arms: TEP hernioplasty

SUMMARY:
This randomized study compares open inguinal hernia repair (Lichtenstein hernioplasty) to endoscopic repair (TEP) in terms of chronic pain and recurrences in one and five years after operation.

DETAILED DESCRIPTION:
The best operative technique in female inguinal hernia is not known. Some register studies recommend always laparoscopic hernia repair in females, but there are no randomized studies to show that laparoscopic repair is better than open hernioplasty. Our study compares operative complications, chronic pain and recurrences in Lichtenstein operation to totally endoscopic hernia repair (TEP) in 170 female patients with primary inguinal hernia. The patients are operated in six Finnish hospitals, randomized into 85 Lichtenstein vs 85 TEP and followed 1 week, 4 weeks, 12 months and 5 years. Main end-point in postoperative pain after one year, sencondary endpoints are sick leave, return to normal physical activity, complications of treatment, re-operations, chronic pain and costs of treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal hernia in females

Exclusion Criteria:

* emergency operation
* recurrent hernia
* groin pain without hernia
* frail and sick patient ASA ≥ 4

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study includes only females
Enrollment: 170 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic pain | from 1 week to one year
  Postoperative inguinal pain (vas scores 0-10) after 1 week, 4 weeks and one year of surgery

SECONDARY OUTCOMES:
Complications | 1 month
  Postoperative complications of surgery (wound infection, hemorrhage)
Recurrence | 5 years
  Hernia recurrences after 5 years
Sick leave | 0-30 days
  how many days the patient is not working after surgery
Treatment costs | 0-30 days
  how much in euros the surgical treatment will cost

CONTACTS AND LOCATIONS:
Locations (1):
- Mikkeli Central Hospital, Mikkeli, Finland

IPD SHARING:
Plan to Share IPD: No